CLINICAL TRIAL: NCT07392242
Title: A Phase II Study of IDH1 Inhibition With Ivosidenib as Maintenance Therapy After Ivosidenib, Azacitidine, and Venetoclax for Acute Myeloid Leukemia
Brief Title: A Study of the Combination of Ivosidenib, Azacitidine, and Venetoclax Followed by Ivosidenib Alone in People With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Servier Pharmaceuticals, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-224
Record Dates: First submitted 2026-01-27; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: Ivosidenib; Azacitidine; Venetoclax; 25-224
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — ivosidenib; Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: This is a phase II, single-arm, multicenter clinical trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivosidenib, Azacitidine, and Venetoclax Followed by Ivosidenib Alone (Experimental): Patients will be initially treated with 7 days of azacitidine (IV or SC per institutional preference, 14 days of venetoclax and 14 days of Ivosidenib daily, days 15 through 28 for cycle 1, then days 1 through 28 for each cycle thereafter).
  Interventions: Drug: Ivosidenib; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Ivosidenib — Ivosidenib ( days 15 through 28 for cycle 1, then days 1 through 28 for each cycle thereafter)
Drug: Azacitidine — Azacitidine (IV or SC per institutional preference, days 1 through 7)
Drug: Venetoclax — Venetoclax (days 1 through 14)

SUMMARY:
The researchers are doing this study to find out whether a 3-drug combination of ivosidenib, azacitidine, and venetoclax followed by maintenance therapy with ivosidenib alone is an effective treatment approach for people with newly diagnosed acute myeloid leukemia (AML) that has an IDH mutation. Maintenance therapy is additional treatment given to help keep cancer from coming back after it has disappeared following the first course of treatment. The researchers will also look at the safety of the treatment approach and what kind of a time commitment it involves for participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 60 years of age at the time of signing the informed consent form (ICF).
* Participant is willing and able to adhere to the study visit schedule and other protocol requirements.
* Participant has newly diagnosed AML as per World Health Organization 2022 or European leukemia Network 2022 guidelines.
* Participant has IDH1-R132 mutation present prior to initiating Ivo/Aza/Ven confirmed by CLIA approved local testing via next-generation sequencing (NGS) and/or polymerase chain reaction (PCR). Other 2-HG producing IDH1 variants may be eligible after discussion with MSK principal investigator.

  1. At MSK, this testing will utilize the MSK-REACT, a rapid multi-gene NGS panel used in all new AML diagnoses that is clinically validated by the Laboratory of Diagnostic Molecular Pathology pursuant to the requirements of CLIA'88 and approved by New York State. Other sites may use local CLIA-certified laboratories and validated clinical assays as per standard of care.
  2. The patient's chart will be utilized for screening purposes
* Participant has Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Participant must have a WBC count <25,000/μL at the time of initiation of study drug (leukapheresis may be performed and/or hydroxyurea may be administered to decrease the WBC count to <25,000/μL).
* Participant has adequate organ function defined as:

  1. Serum aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 3 x ULN, unless considered due to leukemic organ involvement.
  2. Serum total bilirubin < 3.0 x ULN. Higher levels are acceptable if these can be attributed to ineffective erythropoiesis, leukemia organ involvement or Gilbert's syndrome.
  3. Serum creatinine < 2 x ULN or creatinine clearance 30 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR) estimation.

Exclusion Criteria:

* Participant with acute promyelocytic leukemia
* Participants who have previously received ivosidenib or venetoclax
* Participant receiving any other investigational anti-cancer agents. Cytoreductive therapy such as hydroxyurea is permitted.
* Participants with immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
* Participant has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
* Participants who are planned for allogeneic stem cell transplantation based on the assessment of the treating clinician.
* Participant has significant active cardiac disease within 6 months prior to start of study treatment, including New York Heart Association (NYHA) class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke
* Participant has active viral infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV). As per exclusion criteria 5, patients receiving appropriate treatment would only be excluded if there is no improvement.
* Participant is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* Participant has QTc interval (i.e., Fridericia's correction [QTcF]) ≥ 450 ms (mean of triplicate ECG) or other factors that increase the risk of QT prolongation or ventricular arrhythmic events (e.g. family history of long QT interval syndrome). Participants with a QTcF over 450 ms due
* Male or female participants not willing to comply with contraceptive requirements

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 12 months
  Event-free survival is defined as the time between date of treatment start to treatment failure (failure to achieve complete remission or <5% bone marrow blasts), confirmed relapse or death.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Kai Chin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/